CLINICAL TRIAL: NCT05218941
Title: New IMPLANTARY SURGERY Protocol ASSISTED BY PASSIVE ROBOTIQUE: Pilot Study
Acronym: NAVIMPLANT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Departure of the principal investigator
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC31/16/8764
Record Dates: First submitted 2022-01-19; First posted 2022-02-01 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Dental Implants
Keywords: implantology; computer aided surgery; control navigation; X-Guide®

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Passive robotic group (Experimental): Implant surgery without flap assisted by passive robotics
  Interventions: Procedure: Implant surgery assisted by passive robotics
- Control group (Active Comparator): Implant surgery with flap
  Interventions: Procedure: Conventional implant surgery

INTERVENTIONS:
Procedure: Implant surgery assisted by passive robotics — Implant surgery without flap assisted by passive robotics (X-Guide®)
  Arms: Passive robotic group
Procedure: Conventional implant surgery — Flap implant surgery
  Arms: Control group

SUMMARY:
The use of a passive robotic system allows the practitioner to widen the field of indications of flapless surgical access to the implant with an increased operative security and the possibility of an operative modification of the surgical protocol.

DETAILED DESCRIPTION:
In recent decades, the placement of dental implants has become a common procedure for the rehabilitation of partially or completely edentulous patients. The placement of implants requires good visibility of the bone support to avoid accidents such as bone fenestration. This is why, except in very favourable cases where the bone crest is wide, unconcavated and with an ideal periodontal support, it was until then necessary to proceed with a flap before placing the implant. This invasive surgical protocol necessary for implant placement with good visual access has negative parameters such as :

* detachment of the periosteum and therefore risk of bone resorption
* longer intervention time
* need for sutures
* post-operative pain. On the other hand, flapless techniques, which respect the periosteum and periodontium, offer simpler surgical outcomes, reduced risk of bleeding and infection, less bone resorption, and overall better healing. However, the absence of an access flap to the implant site requires special anatomical conditions to avoid any risk of bone fenestration during drilling, and this technique is directly related to the operator's experience. Increasing the number of cases treated by flap-free implant surgery with increased safety is now possible thanks to computer-assisted surgery and passive robotics.

The main objective is to compare the patient's post-operative pain outcomes between passive robotic implant surgery and conventional implant surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 21 years old
* Favorable diagnosis of implant placement regardless of technique (ambivalence clause)
* Radiological situation with sufficient bone volume but requiring a muco-gingival flap or the help of passive robotics.
* Affiliated or beneficiary of a social security
* Signed informed consent

Exclusion Criteria:

* Patient eligible for one or more implants and having a broad bone crest, with no marked concavity, and covered with a sufficient amount of keratinized attached gum.
* Patient with limited oral opening
* Patient with contraindications to implant placement (valve prostheses, unbalanced diabetes)
* Photosensitive epileptic patient
* Patient refusal to participate in the study
* Pregnant or breastfeeding woman
* Patients under guardianship or curatorship

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Pain assessment | 24 hours
  Pain assessment according to a visual analogue scale ranging from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Antoine GALIBOURG, Principal Investigator — galibourg.a@chu-toulouse.fr
Locations (1):
- Toulouse University Hospital, Toulouse, France